CLINICAL TRIAL: NCT01728207
Title: A Phase I Dose Escalation Study of Immunotherapy With IMMU-114 in Patients With Non-Hodgkin's Lymphoma (NHL) and Chronic Lymphocytic Leukemia (CLL)
Brief Title: Phase I Dose Escalation Study of IMMU-114 in Relapsed or Refractory NHL and CLL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was stopped due to insufficient efficacy and very slow accrual
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMMU-114-01
Record Dates: First submitted 2012-11-13; First posted 2012-11-19 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2020-03

CONDITIONS: Non-hodgkin's Lymphoma; Follicular Lymphoma; Mantle Cell Lymphoma; Marginal Zone Lymphoma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: NHL; CLL; follicular lymphoma; mantle cell lymphoma; marginal zone lymphoma; chronic lymphocytic leukemia; small lymphocytic lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — IMMU-114

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMMU-114 (Experimental): IMMU-114 will be administered subcutaneously (under the skin) once or twice weekly for 3 weeks followed by one week of rest. Treatment cycles will continue until disease worsening or toxicity. Various dose levels will be studied.
  Interventions: Drug: IMMU-114

INTERVENTIONS:
Drug: IMMU-114 — hL243 is a humanized antibody that targets HLA-DR, which is found on various b-cell hematologic malignancies and in autoimmune diseases.
  Other Names: hL243

SUMMARY:
IMMU-114 will be studied at different dose schedules and dose levels in order to assess the highest dose safely tolerated. IMMU-114 will be administered subcutaneously (under the skin). IMMU-114 will be given 1-2 times weekly for 3 weeks followed by one week of rest. This is considered one cycle. Treatment cycles will be repeated until toxicity or worsening of disease.

ELIGIBILITY:
Inclusion Criteria:

* Each patient with CLL/SLL must meet all of the following inclusion criteria to be enrolled on the study:
* Patients must have met the diagnostic criteria for CLL/SLL according to the IWCLL 2008 [13] or WHO Guidelines at some point during their disease course:
* Patients with SLL: tumor biopsy immunohistochemistry diagnostic of SLL or blood/bone marrow immunophenotype similar to CLL without lymphocytosis and enlarged lymph nodes.
* Patient must have relapsed or refractory CLL/SLL following at least one purine analog-containing regimen (or after one non-purine analog containing regimen if there is a relative contraindication to purine-analog containing therapy) and not have traditional options available or decline these. Patients with prolymphocytic leukemia (PLL)-CLL or PLL transformation of CLL are eligible.
* Patients must meet IWCLL 2008 Guideline [13] criteria for active disease requiring treatment.

Each patient with NHL must meet all of the following inclusion criteria to be enrolled on the study:

* Patients with histologically confirmed B-cell NHL including marginal zone lymphoma, follicular lymphoma, or mantle cell lymphoma by WHO criteria.
* Patients must have relapsed or refractory disease after at least one prior therapy and not have traditional options available or decline these.

All patients must meet all of the following inclusion criteria to be enrolled on the study:

* Age ≥ 18 years
* Able to understand and sign a written informed consent document.
* Able to receive outpatient treatment and follow-up at the treating institution.
* ECOG performance status 0-1.
* Relapsed/refractory to at least one prior standard systemic treatment regimen, but no more than 4.
* Completed all prior therapies (immunosuppressive medications, antineoplastic therapy, vaccination, immunotherapy, chemotherapy, radiotherapy, major surgery, etc) >4 weeks prior to the first study dose of medication (alemtuzumab ≥ 6 months).
* If receiving corticosteroids, ≤ 20 mg/day prednisone or equivalent and unchanged
* Patients capable of reproduction and male patients who have partners capable of reproduction must agree to use an effective contraceptive method during the course of the study and for 2 months following the completion of their last treatment.
* Females of childbearing potential must have a negative serum β-Hcg pregnancy test result within 7 days of first study dose. Female patients who are surgically sterilized or who are > 45 years old and have not experienced menses for > 2 years may have β- Hcg pregnancy test waived.
* Required baseline laboratory data
* Platelet count ≥ 75,000/mm3
* Absolute neutrophil count (ANC) ≥ 1500/mm3
* AST/ALT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine and total bilirubin ≤ 1.5 times ULN

Exclusion Criteria:

* Patients having received anti-CD20 therapy ≤ 4 weeks prior to the first study dose.
* Patients having received alemtuzumab (anti-CD52) therapy ≤ 6 months prior to the first study dose.
* Patients having undergone prior allogeneic stem cell transplantation within 6 months or having active graft versus host disease.
* Patients with active Richter's syndrome (>10% large B-cells in marrow).
* Patients that have been designated Class III or IV by the New York Heart Association Functional Classification.
* Patients with a history of myocardial infarction or stroke within the last 6 months
* Patients with transfusion-dependent anemia.
* Patients with known hypersensitivity to any excipient contained in the drug formulation.
* Patients with a history of documented human anti-globulin antibodies.
* Patients with active viral, bacterial or systemic fungal infection requiring treatment.
* Patients who are known to be HIV or hepatitis C positive.
* Patients with a history of prior secondary malignancy that requires active systemic therapy that will interfere with interpretation of efficacy or toxicity of IMMU-114, or limit survival to 2 years. These patients should be discussed with the sponsor prior to enrollment. Patients with basal or squamous skin carcinoma, cervical carcinoma in situ on biopsy, localized breast cancer requiring hormonal therapy or localized prostate cancer (Gleason score < 5) do not require discussion.
* Patients with active known CNS lymphoma. Patients with history of CNS leukemia now in remission are eligible for the trial.
* Patients who are pregnant or breast-feeding.
* Patients with major surgery or radiation therapy within 4 weeks prior to first study dose.
* Patients must have recovered all toxicities from prior therapy or radiation to grade 1 or less (excluding alopecia).
* Patients with substance abuse or other medical or psychiatric conditions that, in the opinion of the investigator, would confound study interpretation or affect the patient's ability to tolerate or complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | Safety will be assessed by measuring the change from baseline during treatment and up to 30 days after treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Clinical Response: o Measured by International Working Group Criteria for NHL patients. o Measured by IWCLL 2008 Guidelines for CLL patients. | Efficacy will be assessed every 12 weeks during treatment and 4 weeks after the end of treatment
  Responders will be defined as those with complete response (CR) or partial response (PR). Overall response rate (ORR) will be calculated as the number of evaluable responders divided by the total number of evaluable patients.
Progression Free Survival | During treatment and the changes at 4, 8 and 12 weeks after treatment and then every 3 months for up to 2 years
Overall Survival | During treatment and the changes at 4, 8 and 12 weeks after treatment and then every 3 months for up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: William Wegener, MD, PhD, Study Chair — Gilead Sciences
Locations (5):
- United States (5):
  - Helen F Graham Cancer Center, Newark, Delaware
  - Nancy N. and J.C. Lewis Cancer and Research Pavilion, Savannah, Georgia
  - Indiana University Health Goshen Hospital, Goshen, Indiana
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Huntsman Cancer Institute, Univ. Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Park KH, Sawada T, Murakami T, Ishii Y, Yasuo M, Fuchinoue S, Goldenberg DM, Kubota K. Anti-class II -DR humanized monoclonal antibody, IMMU-114, blocks allogeneic immune response. Am J Surg. 2012 Oct;204(4):527-34. doi: 10.1016/j.amjsurg.2011.11.017. Epub 2012 Jun 1. PMID 22658578
- [Background] Chen X, Chang CH, Stein R, Goldenberg DM. The humanized anti-HLA-DR moAb, IMMU-114, depletes APCs and reduces alloreactive T cells: implications for preventing GVHD. Bone Marrow Transplant. 2012 Jul;47(7):967-80. doi: 10.1038/bmt.2011.203. Epub 2011 Oct 24. PMID 22020022
- [Background] Rossi EA, Rossi DL, Cardillo TM, Stein R, Goldenberg DM, Chang CH. Preclinical studies on targeted delivery of multiple IFNalpha2b to HLA-DR in diverse hematologic cancers. Blood. 2011 Aug 18;118(7):1877-84. doi: 10.1182/blood-2011-03-343145. Epub 2011 Jun 16. PMID 21680794
- [Background] Stein R, Balkman C, Chen S, Rassnick K, McEntee M, Page R, Goldenberg DM. Evaluation of anti-human leukocyte antigen-DR monoclonal antibody therapy in spontaneous canine lymphoma. Leuk Lymphoma. 2011 Feb;52(2):273-84. doi: 10.3109/10428194.2010.535182. Epub 2010 Dec 6. PMID 21133722
- [Background] Stein R, Gupta P, Chen X, Cardillo TM, Furman RR, Chen S, Chang CH, Goldenberg DM. Therapy of B-cell malignancies by anti-HLA-DR humanized monoclonal antibody, IMMU-114, is mediated through hyperactivation of ERK and JNK MAP kinase signaling pathways. Blood. 2010 Jun 24;115(25):5180-90. doi: 10.1182/blood-2009-06-228288. Epub 2010 Jan 25. PMID 20101022